CLINICAL TRIAL: NCT00774319
Title: A Randomised Study of TPF as Neoadjuvant Chemotherapy Followed by Concomitant Chemoradiotherapy (CRT) With Conventional Radiotherapy (RT) Versus Concomitant CRT With Accelerated RT in Patients With Locally Advanced Head and Neck Squamous Cell Cancer (HNSCC) in Good Condition. The Condor Study. A Study of the Dutch Head and Neck Cancer Group (DHNCG).
Brief Title: TPF Induction With Concomitant Chemoradiation to Treat Patients With Head and Neck Cancer
Acronym: Condor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NWHHT08-01
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Head and Neck Cancer
Keywords: HNSCC; neo Adjuvant; Chemoradiation therapy; TPF
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Induction Chemotherapy with TPF Then: cisplatin 100 mg/m2 on day 1, 22 and 43 combined with conventional radiotherapy
  Interventions: Radiation: conventional radiotherapy with 'high' dose cisplatin
- 2 (Active Comparator): Induction chemotherapy with TPF Then cisplatin 40mg/m2 on day 1,8,15,22,29 and 35 combined with accelerated radiotherapy
  Interventions: Radiation: accelerated radiotherapy with 'low' dose cisplatin

INTERVENTIONS:
Radiation: conventional radiotherapy with 'high' dose cisplatin — radiotherapy: 5 fractions/week, total treatment time 7 weeks. Dose to gross tumor volume 70 Gy/35 fractions, dose to elective nodal areas 46 Gy/23 fractions.
  100 mg/m2 cisplatin iv on day 1, 22 and 43
  Arms: 1
Radiation: accelerated radiotherapy with 'low' dose cisplatin — Accelerated radiotherapy 6 fractions/week, total treatment time 6 weeks. During one of the weekdays two fractions will be delivered with an interval of at least 6h. Dose to gross tumor volume 70 Gy/35 fractions, dose to elective nodal areas 46 Gy/23 fractions cisplatin 40 mg/m2 iv on day 1,8,18,22,29,35
  Arms: 2

SUMMARY:
The purpose of this trial is to compare two different treatments for fit patients with head and neck cancer:

All patients are given induction-chemotherapy (docetaxel, cisplatin, 5-FU).

Subsequently patients are being randomised into two groups:

* The first group receives neo-adjuvant chemotherapy ('high' dose cisplatin) and conventional radiotherapy
* The second group receives neo-adjuvant chemotherapy ('low' dose cisplatin) and accelerated radiotherapy.

DETAILED DESCRIPTION:
Induction Chemotherapy TPF(arm A and B)

: Docetaxel 75 mg/m2 iv on day 1, Cisplatin 75 mg/ m2 iv on day 1, 5-FU 750 mg/ m2/day iv continuous infusion (in Hickman or port a cath) on days 1-5; prophylactic G-CSF

This cycle will be repeated every 21 days for a maximum of 4 cycles. Clinical evaluation after each cycle and radiological evaluation after 2 cycles will take place. In case of PD or SD (after 2 cycles) with no minor response (no decrease in measurable disease from baseline) concomitant chemoradiotherapy will started per protocol.

Surgery The investigators in each centre can decide neck surgery for residual tumor

ELIGIBILITY:
Inclusion Criteria:

Histology and staging disease

* Histologically or cytologically proven non-metastatic locally advanced HNSCC, stage III or IV, for which concomitant chemo-radiotherapy would be the standard therapy
* Patients can be included either with irresectable disease or for which the concomitant chemoradiotherapy was chosen for organ preservation
* Measurable disease
* Primary site: oral cavity, oropharynx, hypopharynx and larynx

General conditions

* Written informed consent
* Age >18 years and ≤ 65 years
* WHO performance status 0-1
* Adequate bone marrow function (WBC > 3.0 x 109/L, platelets > 100 x 109/L, Hb > 6 mmol/L)
* Adequate hepatic function: total bilirubin < 1. 5 x upper normal limit, ASAT and ALAT < 2.5 x upper normal limits
* Adequate renal function: calculated creatinin clearance > 60ml/min. (Cockcroft-Gault formula) Other
* Expected adequacy of follow-up.

Exclusion Criteria:

General conditions

* Active alcohol addiction
* Admission for COPD in the last 12 months
* Weight loss > 10% in 3 months before entry
* Pregnancy or lactation
* Patients (M/F) with reproductive potential not implementing adequate contraceptives measures

Prior or current history

* Prior surgery, radiotherapy or chemotherapy for this tumor
* Serious concomitant diseases preventing the safe administration of chemotherapy and/or radiotherapy or likely to interfere with the study assessments
* Serious active infections
* Other malignancies in the past 5 years with the exception of adequately treated carcinoma in situ of the cervix, or squamous or basal cell carcinoma of the skin

Concomitant treatments

* Concomitant (or within 4 weeks before randomisation) administration of any other experimental drug under investigation
* Concurrent treatment with any other anti-cancer therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2008-12; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
feasibility of both study-arms | 2 years

SECONDARY OUTCOMES:
to assess the toxicity profile, tumour response, disease free survival and overall survival in both study-arms. Also QoL will be measured. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: C.M.L. van Herpen, MD, Phd, Principal Investigator — UMCN st Radboud
Locations (2):
- Netherlands (2):
  - Netherlands Cancer Institute, Amsterdam
  - University Medical Center Nijmegen st Radboud, Nijmegen

REFERENCES:
- [Derived] Driessen CML, Groenewoud JMM, de Boer JP, Gelderblom H, van der Graaf WTA, Prins JB, Kaanders JHAM, van Herpen CML. Quality of life of patients with locally advanced head and neck cancer treated with induction chemotherapy followed by cisplatin-containing chemoradiotherapy in the Dutch CONDOR study: a randomized controlled trial. Support Care Cancer. 2018 Apr;26(4):1233-1242. doi: 10.1007/s00520-017-3946-7. Epub 2017 Dec 11. PMID 29230548
- [Derived] Driessen CM, de Boer JP, Gelderblom H, Rasch CR, de Jong MA, Verbist BM, Melchers WJ, Tesselaar ME, van der Graaf WT, Kaanders JH, van Herpen CM. Induction chemotherapy with docetaxel/cisplatin/5-fluorouracil followed by randomization to two cisplatin-based concomitant chemoradiotherapy schedules in patients with locally advanced head and neck cancer (CONDOR study) (Dutch Head and Neck Society 08-01): A randomized phase II study. Eur J Cancer. 2016 Jan;52:77-84. doi: 10.1016/j.ejca.2015.09.024. Epub 2015 Dec 1. PMID 26655558